CLINICAL TRIAL: NCT03570970
Title: Multiple-dose Tolerability and Pharmacokinetic Studies of Benapenem for Injection in Phase Ib Clinical Healthy Subjects
Brief Title: Multiple-dose Tolerability and Pharmacokinetic Studies of Benapenem inClinical Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sihuan Pharmaceutical Holdings Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5081-CPK-1003
Record Dates: First submitted 2018-05-17; First posted 2018-06-27 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-05

CONDITIONS: Healthy Subject

STUDY DESIGN:
Intervention Model Description: 250 mg group is performed firstly. After completion of observation and confirming that the drug can be safely tolerated, study on 500 mg group is then performed. After completion of observation and confirming that the drug can be safely tolerated, study on 1000 mg group is then performed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Banapenem C1 group (Experimental): 250mg Once daily for 7
  Interventions: Drug: Banapenem
- Banapenem C2group (Experimental): 500mg Once daily for 7
  Interventions: Drug: Banapenem
- Banapenem C3group (Experimental): 1000mg Once daily for 7
  Interventions: Drug: Banapenem

INTERVENTIONS:
Drug: Banapenem — Banapenem to be used anti-infection
  Other Names: 5081

SUMMARY:
To observe the pharmacokinetic profiles of benapenem and its major metabolites in healthy volunteers after continuous multiple-dose benapenem, providing evidence for phase Ⅱ clinical study.

DETAILED DESCRIPTION:
A single-center, randomized, open-label, and dose escalation trial design is used in the multiple-dose tolerability and pharmacokinetic studies. The tolerability and pharmacokinetic studies are performed simultaneously. Three doses, 250 mg, 500 mg, and 1000 mg are proposed for multiple-dose tolerability and pharmacokinetic studies. The subjects are divided into two groups, 12 subjects in each group, half males and half females. 250 mg group is performed firstly. After completion of observation and confirming that the drug can be safely tolerated, study on 500 mg group is then performed. After completion of observation and confirming that the drug can be safely tolerated, study on 1000 mg group is then performed. Each subject only receives one dose, intravenous drip, once daily, for 7 consecutive days. During the trial, close attention is paid to the tolerability of subjects, and blood samples 4 mL is collected from cubital vein respectively before dosing, 0.25 h, 0.5 h, 0.75 h, 1 h, 1.5 h, 2 h, 3 h, 5h, 8 h, 12 h, and 24 h after dosing on Day 1 (0 h); before dosing (0 h), 0.25 h, 0.5 h, 0.75 h, 1 h, 1.5 h, 2 h, 3 h, 5 h, 8 h, 12 h, 24 h, 36 h, and 48 h after dosing on Day 7 for pharmacokinetic study. Blood samples are collected before dosing on Day 4, 5 and 6 to determine the trough concentration for observing the pharmacokinetic profiles of benapenem and its major metabolites in the body after continuous dosing. The next dose group can be studied only when the observation of the previous dose group is completed and it is confirmed that the drug is safely tolerated

ELIGIBILITY:
Inclusion Criteria:

* Male or female healthy subjects, aged 18~45;
* Body weight ≥ 50 kg and body mass index 19.0~24.0 kg/m2;
* To the test, physical examination, blood routine, urine routine, liver and kidney functions, and related examinations normal, or mild abnormalities in indicators while without clinical significance as indicated by the investigator;
* Normal or mild abnormalities without clinical significance in the standard 12-lead ECG;
* Signing informed consent form.

Exclusion Criteria:

* Regular smoking, alcohol abuse, and drug abuse;
* Use of drugs with known damage to an organ within three months;
* History of specific allergies , or history of drug allergy, especially those allergic to lactams and excipients of test drug;
* Febrile illnesses within three days before the screening;
* Patients with mental illness or psychotic disorder in the past;
* Past nervous system diseases (epilepsy, stroke, cerebrovascular disorder, etc.), gastrointestinal disorder (such as stomach ulcers, gastritis, etc.) or disorder of other systems (such as cardiovascular, respiratory, hematological, or endocrine system, etc.) diseases or medical history.
* Habitually taking any medication, including traditional Chinese medicine;
* Having taken any medication that may affect test results within two weeks before the screening, such as antibiotics, NSAIDs, aluminum- or magnesium-containing antacids, diuretics, anticoagulants, central nervous system depressants, and any drug that may affect the drug absorption;
* Having participated in other investigational drug trial in the preceding three months;
* Blood donation for 360 ml or more within three months before the screening;
* Heart rate<50bpm or >100bpm; 12)Systolic blood pressure <90 mmHg or ≥140 mmHg, diastolic blood pressure ≥90mmHg or <60mmHg;
* Women who are pregnant or breastfeeding, or who may be pregnant without adopting acceptable contraception, or who have a positive result in serum pregnancy test;
* Women who are planning to become pregnant within 6 months, or male subjects who are planning to make his spouse pregnant within 6 months;
* HBsAg, HCV antibody, HIV antibody, and Treponema pallidum antibody positive;
* Urine drug-of-abuse testing positive;
* Any other factor that makes the subject not suitable for the trial as indicated by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-03-14 (Actual); Primary Completion 2016-06-02 (Actual); Study Completion 2016-06-02 (Actual)

PRIMARY OUTCOMES:
AUC(0-24) of Benapenem | Pre dose and 0.25,0.5,0.75,1,1.5, 2, 2.5, 3, 4, 6,8,12, 24hours after Dosing
  AUC(0-24) is the area under the curve from time 0 to 24 hour
Maximum observed plasma concentration (Cmax) of Benapenem | Pre dose and 0.25,0.5,0.75,1,1.5, 2, 2.5, 3, 4, 6,8,12, 24hours after Dosing
  Maximum observed plasma concentration (Cmax) of Benapenem in healthy subjects
Time to maximum observed plasma concentration (tmax) of Benapenem | Pre dose and 0.25,0.5,0.75,1,1.5, 2, 2.5, 3, 4, 6,8,12, 24hours after Dosing
  Time to maximum observed plasma concentration (tmax) of Benapenem in healthy subjects
Time to elimination half-life (t1/2) of Benapenem | Pre dose and 0.25,0.5,0.75,1,1.5, 2, 2.5, 3, 4, 6,8,12, 24hours after Dosing
  Time to elimination half-life (t1/2) of Benapenem in healthy subjects

SECONDARY OUTCOMES:
Number of subjects with clinically significant findings in vital signs | Screening, Day1, Day2, Day4 after Dosing
  Vitals signs such as systolic and diastolic blood pressure, heart rate, and pulse rate will be measured in a semi-supine position after 5 minutes of rest
Number of subjects with clinically significant findings in laboratory parameters | Screening, Day1, Day2, Day4 after Dosing
  Hematology and Clinical Chemistry and Urine routine abnormalities will be monitored
Number of subjects with clinically significant 12-lead ECGs | Screening, Day1, Day2, Day4 after Dosing
  Single 12-lead ECGs will be obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTcF intervals.
Number of subjects with adverse events and serious adverse events | From Screening to Day 4 after dosing
  All adverse events will be monitored in each group subjects

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Lv, PhD, Principal Investigator — Peking University First Hospital

REFERENCES:
- [Derived] Zhao CY, Lv Y, Zhu Y, Wei MJ, Liu MY, Ji XW, Kang ZS, Xia YH, Tian JH, Ma Y, Liu Y. A First-in-Human Safety, Tolerability, and Pharmacokinetics Study of Benapenem in Healthy Chinese Volunteers. Antimicrob Agents Chemother. 2019 Feb 26;63(3):e02188-18. doi: 10.1128/AAC.02188-18. Print 2019 Mar. PMID 30617093